CLINICAL TRIAL: NCT05406648
Title: The Effect of Black Mulberry (Morus Nigra) Consumption on Cognitive Functions and Antioxidant Capacity in Individuals Diagnosed With Dementia
Brief Title: The Effect of Black Mulberry (Morus Nigra) Consumption on Cognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Yuksek Ihtisas University (Other); Gulhane Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeynep Goktas, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-AKD-167
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 20g of Morus nigra concentrate administration for 12 weeks
  Interventions: Other: Morus nigra concentrate
- Control (No Intervention): No intervention throughout the study

INTERVENTIONS:
Other: Morus nigra concentrate — The experimental group was given 20 grams of black mulberry (morus nigra) concentrate per day for 12 weeks.
  Arms: Intervention

SUMMARY:
The study was conducted with 44 patients who were diagnosed with mild-to-moderate Alzheimer's Disease. Participants were divided into 2 groups intervention group and the control group. The intervention group was administered 20 grams of black mulberry concentrate per day for 12 weeks and the control group received no intervention thorough the study. Cognitive functions, antioxidant capacity, and inflammation markers were evaluated at the baseline and at the end of the 12 weeks.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of black mulberry on cognitive functions and biochemical parameters in patients with Alzheimer's disease. The study was conducted in a tertiary geriatric outpatient clinic with 44 patients aged over 65 years who were diagnosed with mild-to-moderate AD. The study was completed by 20 participants in the intervention group and 19 participants in the control group. The intervention group was administered 20 grams of black mulberry concentrate per day for 12 weeks. There was no intervention in the control group (n=19). Routine medical treatment for all participants was continued throughout the study. During the evaluation of the cognitive situation, Mini-Mental State Assessment (MMSA) and AD Assessment Scale-Cognitive Subscale (ADAS-Cog) test were administered. Geriatric Depression Scale (GDS-15) was used to screen for depression symptoms. In order to evaluate antioxidant capacity in serum samples Superoxide dismutase (SOD) enzyme, Total Oxidant Status (TOS), Total Antioxidant Status (TAS), and oxidative stress index level were examined. Furthermore, in order to evaluate lipid oxidation, Malondialdehyde (MDA) level was examined. For the evaluation of inflammation, serum Interleukin 1-beta (IL-1 beta) and Transforming growth factor-beta (TGF-beta) levels were measured.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with dementia in the first stage
* To be using the same medication for dementia throughout the study
* To have been taking the same dementia medication for the last 6 months and no dose changes for at least 3 months
* Not to have used anthocyanin supplement regularly in the last four months before participating in the study
* Confirmation of medication use by caregivers
* To have a caregiver to follow the patient's daily intake of black mulberry concentrate

Exclusion Criteria:

* Those under 65 years of age
* Those who have taken new dementia medication in the last 3 months
* Those staying in nursing homes
* Those with mild cognitive impairment who have not yet been diagnosed with dementia
* Those who have cancer
* Those with inflammatory diseases (viral or bacterial)
* History of head trauma that may lead to unconsciousness or other neurological diseases other than dementia
* Those with a defined autoimmune disease
* Alcohol and drug addiction
* Those with major depression
* Those with uncontrollable hypertension
* Those with uncontrolled diabetes
* Those with dysphagia
* Tube fed
* Those who are bedridden
* Delirium
* Those who use drugs that may affect outcome measures, such as benzodiazepines
* Due to the risk that black mulberry may cause possible food-drug interaction via p-glycoprotein / CYP3A in the literature, patients using the drugs named below will not be included in the study.

  1. Antineoplastic drugs (docetaxel, etoposide, vincristine),
  2. Calcium channel blockers (eg amlodipine)
  3. Calcineurin inhibitors (tacrolimus and cyclosporine)
  4. Digoxin
  5. Macrolide antibiotics (Clarithromycin)
  6. Protease inhibitors

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Change in cognition (ADAS-Cog) | 12 weeks
  Change in Alzheimer's Disease Assessment Scale-Cognitive Subscale scores
Change in cognition (MMSE) | 12 weeks
  Change in Mini-Mental State Examination scores
Antioxidant capacity (TOS) | 12 weeks
  Change in serum Total Oxidant Status (TOS)
Antioxidant capacity (TAS) | 12 weeks
  Change in serum Total Antioxidant Status (TOS)

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Goktas, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No